CLINICAL TRIAL: NCT04988776
Title: Comparison Between Ultrasound-guided Pectoral Nerves Block Type II and Intercostobrachial Nerve Block as a Supplement to Supraclavicular Block for Anesthesia of Proximal Arteriovenous Access in End-stage Renal Disease Patients
Brief Title: PECS II Versus ICBN Block Plus SCNB for AV Fistula Creation in CRF Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Menoufia University (Other)
Collaborators: Mamdoh Elsayed Lotfy (Unknown); amany aly sultan (Unknown); reem gaber abdel-mageed (Unknown)
Responsible Party: Principal Investigator, ashraf magdy eskandr, assistant professor of anesthesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PECS II versus ICBN block
Record Dates: First submitted 2021-07-25; First posted 2021-08-03 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Intraoperative Analgesia; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Active Comparator): Patients received ultrasound-guided Intercostobrachial nerve block with 10 ml 0.25% bupivacaine (5 ml 0.5% bupivacaine will be added to 5ml 0.9% normal saline ) supplemental to supraclavicular block with 30 ml 0.25% bupivacaine (15 ml 0.5% bupivacaine will be added to 15 ml of 0.9 %Nacl ) .
  Interventions: Other: ultrasUltrasound-guided Intercostobrachial nerve block supplemental to supraclavicular block with 30 ml 0.25% bupivacaine (15 ml 0.5% bupivacaine will be added to 15 m
- group B (Active Comparator): patients received ultrasound-guided pectoral nerves block type II with 10 ml 0.25% bupivacaine (5 ml 0.5% bupivacaine will be added to 5ml 0.9% normal saline ) supplemental to supraclavicular block with 30 ml 0.25% bupivacaine (15 ml 0.5% bupivacaine will be added to 15 ml of 0.9 %Nacl )
  Interventions: Other: ultrasound-guided pectoral nerves block type II supplemental to supraclavicular block

INTERVENTIONS:
Other: ultrasUltrasound-guided Intercostobrachial nerve block supplemental to supraclavicular block with 30 ml 0.25% bupivacaine (15 ml 0.5% bupivacaine will be added to 15 m — patients recieved ultrasound-guided Intercostobrachial nerve block with 10 ml 0.25% bupivacaine (5 ml 0.5% bupivacaine will be added to 5ml 0.9% normal saline ) supplemental to supraclavicular block with 30 ml 0.25% bupivacaine (15 ml 0.5% bupivacaine will be added to 15 ml of 0.9 %Nacl ) .
  Arms: group A
Other: ultrasound-guided pectoral nerves block type II supplemental to supraclavicular block — Patients received ultrasound-guided pectoral nerves block type II with 10 ml 0.25% bupivacaine (5 ml 0.5% bupivacaine will be added to 5ml 0.9% normal saline ) supplemental to supraclavicular block with 30 ml 0.25% bupivacaine (15 ml 0.5% bupivacaine will be added to 15 ml of 0.9 %Nacl )
  Arms: group B

SUMMARY:
Brachial plexus block (BPB) is often utilized for proximal arm arteriovenous access creation. However, the medial upper arm and axilla are often inadequately anesthetized, as the Intercostobrachial nerve (which provides sensory supply to the axilla, upper medial arm, and a small area at the upper lateral chest) is not a component of the brachial plexus. This requires repeated, an intraoperative local anesthetic (LA) supplementation up to conversion into GA. The intercostobrachial nerve (ICBN) is a purely sensory nerve that arises primarily from the second intercostal nerve (T2) with occasional contribution from T3. Therefore, It is not a component of the brachial plexus and is not anesthetized by brachial plexus blockade. The ICBN can be blocked together with other nerves, such as the pectoral, intercostal, and long thoracic nerves in a recently described technique named pectoral nerves block type II (PECS II ).In this thesis, investigators compared the use of the PECS II block and ICBN block as a supplement to supraclavicular brachial plexus block for providing complete anesthesia of the upper arm for fistula creation surgery.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients.
* Proximal Arm Arteriovenous Access Surgery.
* Elective or emergency surgery
* American Society of Anesthesiology (ASA) physical status II to III.

Exclusion Criteria:

* Inability of the patient to provide informed consent, communicate or cooperate
* History of allergy to local anesthetics.
* Preexisting upper limb neurological disease at the side of the surgery.
* Patients on anticoagulant therapy or with history of coagulopathy.
* Previous surgery at or near the site of the study.
* The presence of skin infection at the puncture site.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
intraoperative local anesthetic requirement | 1-2 hours after surgery start
  volume of local anesthetic

SECONDARY OUTCOMES:
postoperative pain | 24 hours after end of surgery
  Visual analogue score (0-10) where 0=no pain and 10=the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: reem abdel-mageed, MBBCh, Principal Investigator — resident of anesthesia, menoufia university hospitals
Locations (1):
- Ashraf Magdy Eskandr, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available after end of the study
Supporting Information: Study Protocol
Time Frame: for 1 year after the end of the study
Access Criteria: study protocol